CLINICAL TRIAL: NCT03468218
Title: A Phase II Trial of Pembrolizumab and Cabozantinib in Patients With RM SCCHN
Brief Title: Pembrolizumab & Cabozantinib in Patients With Head and Neck Squamous Cell Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Exelixis (Industry); National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Nabil F. Saba, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00100269; NCI-2017-02419 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); Winship4234-17 (Other: Winship Cancer Institute); P30CA138292 (NIH)
Record Dates: First submitted 2018-03-10; First posted 2018-03-16 (Actual); Results first posted 2024-12-27 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Head and Neck Carcinoma; Paranasal Sinus Squamous Cell Carcinoma; Recurrent Head and Neck Squamous Cell Carcinoma; Recurrent Hypopharyngeal Squamous Cell Carcinoma; Recurrent Laryngeal Squamous Cell Carcinoma; Recurrent Oral Cavity Squamous Cell Carcinoma; Recurrent Oropharyngeal Squamous Cell Carcinoma; Stage IV Hypopharyngeal Squamous Cell Carcinoma AJCC v7; Stage IV Laryngeal Squamous Cell Carcinoma AJCC v7; Stage IV Oral Cavity Squamous Cell Carcinoma AJCC v6 and v7; Stage IV Oropharyngeal Squamous Cell Carcinoma AJCC v7; Stage IVA Hypopharyngeal Squamous Cell Carcinoma AJCC v7; Stage IVA Laryngeal Squamous Cell Carcinoma AJCC v7; Stage IVA Oral Cavity Squamous Cell Carcinoma AJCC v6 and v7; Stage IVA Oropharyngeal Squamous Cell Carcinoma AJCC v7; Stage IVB Hypopharyngeal Squamous Cell Carcinoma AJCC v7; Stage IVB Laryngeal Squamous Cell Carcinoma AJCC v7; Stage IVB Oral Cavity Squamous Cell Carcinoma AJCC v6 and v7; Stage IVB Oropharyngeal Squamous Cell Carcinoma AJCC v7; Stage IVC Hypopharyngeal Squamous Cell Carcinoma AJCC v7; Stage IVC Laryngeal Squamous Cell Carcinoma AJCC v7; Stage IVC Oral Cavity Squamous Cell Carcinoma AJCC v6 and v7; Stage IVC Oropharyngeal Squamous Cell Carcinoma AJCC v7; Unresectable Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — cabozantinib; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (pembrolizumab, cabozantinib) (Experimental): Patients receive pembrolizumab IV over 30 minutes on day 1 and cabozantinib PO QD on days 1-21. Cycles repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cabozantinib; Biological: Pembrolizumab

INTERVENTIONS:
Drug: Cabozantinib — Given PO
  Other Names: Cabometyx; Cometriq
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475

SUMMARY:
This phase II trial studies how well pembrolizumab and cabozantinib in treating patients with head and neck squamous cell cancer that has come back or spread to other places in the body and cannot be removed by surgery. Monoclonal antibodies, such as pembrolizumab, may interfere with the ability of tumor cells to grow and spread. Cabozantinib may stop the growth of tumor cells by blocking some of the pathways needed for cell growth. Giving pembrolizumab and cabozantinib may improve the chances of tumor response in patients with head and neck squamous cell cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

To estimate the overall response rate (ORR) of patients with recurrent/metastatic (RM) squamous cell carcinoma of the head and neck (SCCHN) who receive the combination of pembrolizumab and cabozantinib.

SECONDARY OBJECTIVES:

* To estimate the progression-free survival (PFS) of patients treated with the combination of pembrolizumab and cabozantinib.
* To further define the toxicities associated with these regimens in patients with SCCHN.

OUTLINE:

Patients receive pembrolizumab intravenously (IV) over 30 minutes on day 1 and cabozantinib orally (PO) once daily (QD) on days 1-21. Cycles repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* The subject has a histologic or cytologic diagnosis of squamous cell carcinoma of the oral cavity, oropharynx, paranasal sinuses, hypopharynx, nasopharynx, or larynx; squamous cell carcinoma of unknown primary in cervical lymph node can be included only if human papillomavirus (HPV) status is positive
* Patients must have refractory, recurrent or metastatic disease, which is deemed to be inoperable
* In case patients received prior systemic therapy within the definitive or metastatic setting, disease progression must be documented following prior therapy; this can be in the recurrent or metastatic setting or in the concurrent setting
* Measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 as determined by the investigator
* A maximum of one prior radiotherapy regimen, curative or palliative, to the head and neck is allowed; if the radiation is combined with chemotherapy, a minimum of 4 months must elapse between the end of radiotherapy and registration; if the radiation is given alone, a minimum of 8 weeks must elapse between the end of radiotherapy and registration; a minimum of 3 weeks must elapse between prior radiation to other areas and registration; treatment areas should be healed with no sequelae from radiation therapy (RT) that would predispose to fistula formation
* The subject has had an assessment of all known disease sites eg, by computerized tomography (CT) scan, magnetic resonance imaging (MRI), bone scan or positron emission tomography (PET)/CT scan as appropriate, within 28 days before the first dose of cabozantinib
* Life expectancy of greater than 3 months
* The subject has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Recovery to baseline or ≤ grade 1 Common Terminology Criteria for Adverse Events (CTCAE) version (v.)4.0 from toxicities related to any prior treatments, unless AE(s) are clinically nonsignificant and/or stable on supportive therapy
* Within 7 days before the first dose of cabozantinib: The absolute neutrophil count (ANC) ≥ 1000/mm³ without colony stimulating factor support
* Within 7 days before the first dose of cabozantinib: Platelets ≥ 100,000/mm³
* Within 7 days before the first dose of cabozantinib: Hemoglobin ≥ 9 g/dL
* Within 7 days before the first dose of cabozantinib: Bilirubin ≤ 1.5 x the upper limit of normal (ULN); for subjects with known Gilbert's disease, bilirubin ≤ 3.0 mg/dL
* Within 7 days before the first dose of cabozantinib: Serum albumin ≥ 2.8 g/dl
* Within 7 days before the first dose of cabozantinib: Serum creatinine ≤ 1.5 x ULN or creatinine clearance (CrCl) ≥ 40 mL/min; for creatinine clearance estimation, the Cockcroft and Gault equation should be used
* Within 7 days before the first dose of cabozantinib: Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.0 x ULN
* Within 7 days before the first dose of cabozantinib: Lipase < 2.0 x the upper limit of normal and no radiologic or clinical evidence of pancreatitis
* Within 7 days before the first dose of cabozantinib: Urine protein/creatinine ratio (UPCR) ≤ 1
* Within 7 days before the first dose of cabozantinib: Serum phosphorus, calcium, magnesium and potassium ≥ lower limit of normal (LLN)
* The subject is capable of understanding and complying with the protocol requirements and has signed the informed consent document
* Sexually active subjects (men and women) must agree to use medically accepted barrier methods of contraception (eg, male or female condom) during the course of the study and for 4 months after the last dose of study drug(s), even if oral contraceptives are also used; all subjects of reproductive potential must agree to use both a barrier method and a second method of birth control during the course of the study and for 4 months after the last dose of study drug(s)
* Female subjects of childbearing potential must not be pregnant at screening; females of childbearing potential are defined as premenopausal females capable of becoming pregnant (ie, females who have had any evidence of menses in the past 12 months, with the exception of those who had prior hysterectomy); however, women who have been amenorrheic for 12 or more months are still considered to be of childbearing potential if the amenorrhea is possibly due to prior chemotherapy, antiestrogens, low body weight, ovarian suppression or other reasons

Exclusion Criteria:

* Patients who have HPV negative squamous cell carcinoma of unknown primary in cervical lymph node
* The subject has received cytotoxic chemotherapy (including investigational cytotoxic chemotherapy) or biologic agents (eg, cytokines or antibodies) within 4 weeks, or nitrosoureas/mitomycin C within 6 weeks before the first dose of study treatment
* Prior treatment with cabozantinib or pembrolizumab
* Radiation therapy for bone metastasis within 2 weeks, any other external radiation therapy within 4 weeks before the first dose of study treatment; systemic treatment with radionuclides within 6 weeks before the first dose of study treatment; subjects with clinically relevant ongoing complications from prior radiation therapy are not eligible
* Receipt of any type of small molecule kinase inhibitor (including investigational kinase inhibitor) within 14 days before the first dose of study treatment
* The subject has received any other type of investigational agent within 28 days or 5 half-lives, whichever is shorter, before the first dose of study treatment
* Known brain metastases or cranial epidural disease unless adequately treated with radiotherapy and/or surgery (including radiosurgery) and stable for at least 4 weeks before the first dose of study treatment; eligible subjects must be neurologically asymptomatic and without corticosteroid treatment at the time of the start of study treatment
* The subject has prothrombin time (PT)/institutional normalized ratio (INR) or partial thromboplastin time (PTT) test ≥ 1.3 x the laboratory ULN within 7 days before the first dose of study treatment
* Concomitant anticoagulation at therapeutic doses with oral anticoagulants (eg, warfarin, direct thrombin and factor Xa inhibitors) or platelet inhibitors (eg, clopidogrel)

  * Note: Low-dose aspirin for cardioprotection (per local applicable guidelines), low-dose warfarin (< 1 mg/day), and low dose, low molecular weight heparins (LMWH) are permitted; anticoagulation with therapeutic doses of LMWH is allowed in subjects who are on a stable dose of LMWH for at least 6 weeks before first dose of study treatment, and who have had no clinically significant hemorrhagic complications from the anticoagulation regimen or the tumor
* The subject has experienced any of the following:

  * Clinically-significant GI bleeding within 6 months before the first dose of study treatment
  * Hemoptysis of ≥ 0.5 teaspoon (2.5 ml) of red blood within 3 months before the first dose of study treatment
  * Any other signs indicative of pulmonary hemorrhage within 3 months before the first dose of study treatment
* The subject has radiographic evidence of cavitating pulmonary lesion(s)
* The subject has tumor invading or encasing any major blood vessels
* The subject has evidence of tumor invading the gastrointestinal (GI) tract (esophagus, stomach, small or large bowel, rectum or anus), or any evidence of endotracheal or endobronchial tumor within 28 days before the first dose of cabozantinib
* The subject has uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

  * Cardiovascular disorders including:

    * Congestive heart failure (CHF): New York Heart Association (NYHA) class III (moderate) or class IV (severe) at the time of screening;
    * Concurrent uncontrolled hypertension defined as sustained blood pressure (BP) > 150 mm Hg systolic or > 100 mm Hg diastolic despite optimal antihypertensive treatment within 7 days of the first dose of study treatment;
    * Any history of congenital long QT syndrome;
    * Any of the following within 6 months before the first dose of study treatment:

      * Unstable angina pectoris;
      * Clinically-significant cardiac arrhythmias;
      * Stroke (including transient ischemic attack (TIA), or other ischemic event);
      * Myocardial infarction;
  * GI disorders particularly those associated with a high risk of perforation or fistula formation including:

    * Tumors invading the GI tract, active peptic ulcer disease, inflammatory bowel disease (eg, Crohn's disease), diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis, acute pancreatitis or acute obstruction of the pancreatic duct or common bile duct, or gastric outlet obstruction
    * Abdominal fistula, GI perforation, bowel obstruction, intra-abdominal abscess within 6 months before randomization

      * Note: Complete healing of an intra-abdominal abscess must be confirmed prior to randomization. Also no pre-existing fistula of head and neck area; no pre-existing osteonecrosis of jaw (ONJ)
  * Other clinically significant disorders that would preclude safe study participation
* Major surgery within 12 weeks before the first dose of study treatment; complete wound healing from major surgery must have occurred 1 month before the first dose of study treatment; minor surgery (including uncomplicated tooth extractions) within 28 days before the first dose of study treatment with complete wound healing at least 10 days before the first dose of study treatment; subjects with clinically relevant ongoing complications from prior surgery are not eligible
* Corrected QT interval by Fridericia's formula (QTcF) > 500 msec within 1 month before the first dose of study treatment

  * Three electrocardiography (ECG)s must be performed for eligibility determination; if the average of these three consecutive results for QTcF is ≤ 500 msec, the subject meets eligibility in this regard
* Pregnant or lactating females
* Inability to swallow intact tablets or inability to take pembrolizumab or cabozantinib
* Previously identified allergy or hypersensitivity to components of the study treatment formulations
* Patients with a history of other prior malignancy must have been treated with curative intent and must have remained disease-free for 1 year post diagnosis; patients with a prior history of squamous cell or basal carcinoma of the skin or in situ cervical cancer must have been curatively treated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-09-18 (Actual); Primary Completion 2022-05-02 (Actual); Study Completion 2026-10-29 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Nabil F. Saba, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia

REFERENCES:
- [Derived] Saba NF, Steuer CE, Ekpenyong A, McCook-Veal A, Magliocca K, Patel M, Schmitt NC, Stokes W, Bates JE, Rudra S, Remick J, McDonald M, Abousaud M, Tan AC, Fadlullah MZH, Chaudhary R, Muzaffar J, Kirtane K, Liu Y, Chen GZ, Shin DM, Teng Y, Chung CH. Pembrolizumab and cabozantinib in recurrent metastatic head and neck squamous cell carcinoma: a phase 2 trial. Nat Med. 2023 Apr;29(4):880-887. doi: 10.1038/s41591-023-02275-x. Epub 2023 Apr 3. PMID 37012550

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Pembrolizumab, Cabozantinib)
Started | 36
Completed | 11
Not Completed | 25
Not completed — Adverse Event | 5
Not completed — Progressive Disease | 16
Not completed — Death | 1
Not completed — Alternate therapy | 1
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Pembrolizumab, Cabozantinib)
Number analyzed (Participants) | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 34
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 27
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 36
Smoking Status [Count of Participants; unit: Participants]
  Current Smoker | 9
  Former Smoker | 8
  Never Smoker | 19

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: Will assess the proportion of subjects with partial response or complete response as defined by Response Evaluation Criteria in Solid Tumors version 1.1 response criteria. ORR will be calculated with 95% confidence interval by binomial distribution. The ability of biomarkers to predict ORR will be estimated by chi-square test and/or logistic regression model.
Time Frame: Up to 2 years after treatment start
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (Pembrolizumab, Cabozantinib)
Number analyzed (Participants) | 36
percentage of participants | 52

2. Secondary Outcome: Progression Free Survival (PFS)
Description: The median PFS will be estimated by Kaplan-Meier method along with 95% confidence interval. The biomarker association with PFS will be assessed by the Kaplan-Meier method, log-rank test, and Cox model.
Time Frame: Duration from date of treatment start to the date of objectively documented progression or death due to any cause, whichever status is recorded first, assessed up to 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Pembrolizumab, Cabozantinib)
Number analyzed (Participants) | 36
percentage of participants | 54 [31.5 to 72]

ADVERSE EVENTS:
Time Frame: 2 years
Description: CTCAE Version 4
Arm/Group | Treatment (Pembrolizumab, Cabozantinib)
All-Cause Mortality (participants affected / at risk) | 7/36
Serious Adverse Events (participants affected / at risk) | 18/36
Other Adverse Events (participants affected / at risk) | 24/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Pembrolizumab, Cabozantinib) (N=36)
Hospitalization-Transanitis (Gastrointestinal disorders) | 1
Hospitalization- Low blood pressure (Vascular disorders) | 1
Hospitalization-hyponatremia (Investigations) | 2
Hospiltaization- acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Hospitalization-drug induced hepatitis (Gastrointestinal disorders) | 1
Death (General disorders) | 7
Hospitalization- Atrial Fibrillation (Cardiac disorders) | 1
Hospitalization-hypotension (Vascular disorders) | 1
Hospitalization- Aspiration (Gastrointestinal disorders) | 2
Hospitalization- Ulcer in right oropharynx (Gastrointestinal disorders) | 1
Hospitalization- Hypercalcemia (Investigations) | 1
Hospitalizaiton- Pancreatitis (Gastrointestinal disorders) | 1
Hospitalization- lower lung consolidation/ NV (Respiratory, thoracic and mediastinal disorders) | 1
Hospitalzation- Leukocytosis, sepsis bowel obstruction (Infections and infestations) | 1
Hospitalizaiton- Anemia (Blood and lymphatic system disorders) | 1
Hospitalization- Back Pain (Musculoskeletal and connective tissue disorders) | 1
Hospitalization- Tachycardia (Cardiac disorders) | 1
Hospitalization- Dysphagia (Gastrointestinal disorders) | 1
Hospitalization- Port infection (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Pembrolizumab, Cabozantinib) (N=36)
Fatigue (General disorders) | 16
Diarrhea (Gastrointestinal disorders) | 13
Hypothyroidism (Endocrine disorders) | 12
Constipation (Gastrointestinal disorders) | 11
Dry Mouth (Gastrointestinal disorders) | 10
Anorexia (Metabolism and nutrition disorders) | 10
Headache (Nervous system disorders) | 10
Hypertension (Vascular disorders) | 12
Hyponatremia (Metabolism and nutrition disorders) | 10
Oral Mucositis (Gastrointestinal disorders) | 9
hypomagnesemia (Metabolism and nutrition disorders) | 8
Pain (General disorders) | 9
Dysphagia (Gastrointestinal disorders) | 10
Hyperglycemia (Metabolism and nutrition disorders) | 8
Palmer-Plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 7
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 8
Abdominal pain (Gastrointestinal disorders) | 6
Back pain (Musculoskeletal and connective tissue disorders) | 8
Hypophosphatemia (Metabolism and nutrition disorders) | 7
Nausea (Gastrointestinal disorders) | 7
Oral Pain (Gastrointestinal disorders) | 7
Maculopapular rash (Skin and subcutaneous tissue disorders) | 6
Decreased white blood count (Blood and lymphatic system disorders) | 6
Anemia (Blood and lymphatic system disorders) | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Dysgeusia (Nervous system disorders) | 5
Respiratory, thoracic and mediastinal disorders-Other, specify (Respiratory, thoracic and mediastinal disorders) | 5
Increased alanine aminotransferase (Metabolism and nutrition disorders) | 5
Increased AST (Metabolism and nutrition disorders) | 6
Dizziness (Nervous system disorders) | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5
Hypotension (Vascular disorders) | 6
Investigations- other (Investigations) | 4
Decreased Platelet Count (Blood and lymphatic system disorders) | 5
Vomiting (Gastrointestinal disorders) | 5
Dehydration (Metabolism and nutrition disorders) | 3
Increased gamma-glutamyl transferase (Hepatobiliary disorders) | 4
General disorders and administration site conditions- Other, specify (General disorders) | 3
Hematuria (Renal and urinary disorders) | 3
Hepatobiliary disorders-Other, specify (Hepatobiliary disorders) | 4
Hypoalbuminemia (Renal and urinary disorders) | 3
Hypocalcemia (Metabolism and nutrition disorders) | 3
Hypokalemia (Metabolism and nutrition disorders) | 3
Increased Lipase (Investigations) | 4
Pain in Extremity (General disorders) | 3
Paresthesia (Nervous system disorders) | 3
acneiform rash (Skin and subcutaneous tissue disorders) | 3
Increased serum amylase (Metabolism and nutrition disorders) | 3
skin and subcutaneous tissue disorders-Other, specify (Skin and subcutaneous tissue disorders) | 3
Weight loss (Gastrointestinal disorders) | 3
Increased alkaline phosphate (Investigations) | 3
Anxiety (Psychiatric disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Aspiration (Respiratory, thoracic and mediastinal disorders) | 3
Increased blood bilirubin (Investigations) | 3
Dry skin (Skin and subcutaneous tissue disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 2
Ear pain (Ear and labyrinth disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Infections and infestations-Other (Infections and infestations) | 2
Leukocytosis (Blood and lymphatic system disorders) | 2
Decreased lymphocyte count (Investigations) | 2
Oral dysesthesia (Gastrointestinal disorders) | 2
Pancreatitis (Hepatobiliary disorders) | 2
Sinusitis (Infections and infestations) | 2
Stomach pain (Gastrointestinal disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
gastric obstruction (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-02-28): https://cdn.clinicaltrials.gov/large-docs/18/NCT03468218/Prot_SAP_001.pdf
  • Informed Consent Form (2022-11-15): https://cdn.clinicaltrials.gov/large-docs/18/NCT03468218/ICF_000.pdf